CLINICAL TRIAL: NCT03333018
Title: Aclidinium Bromide Drug Utilisation Post-Authorisation Safety Studies (DUS): Common Protocol for Aclidinium (DUS1) and Aclidinium/Formoterol Fixed-Dose Combination (DUS2)
Brief Title: A Drug Utilisation Post-authorisation Study of New Users of Aclidinium Bromide (Monotherapy or in Combination)
Acronym: DUS1/DUS2
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: RTI Health Solutions (Other)
Responsible Party: Sponsor
Other Study IDs: D6560R00005; EUPAS6559 (Registry Identifier: ENCePP)
Record Dates: First submitted 2017-10-06; First posted 2017-11-06 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide; Formoterol Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Aclidinium bromide monotherapy: In DUS1, all new users of aclidinium either on monotherapy or with concomitant formoterol will be included. In addition, in DUS2, all new users of the fixed-dose combination of aclidinium/formoterol and any other new fixed-dose combinations of LAMAs and LABAs that become available during the study and that are captured in each database will be included.
  Interventions: Drug: Aclidinium bromide
- Aclidinium bromide and formoterol: In DUS1, all new users of aclidinium either on monotherapy or with concomitant formoterol will be included. In addition, in DUS2, all new users of the fixed-dose combination of aclidinium/formoterol and any other new fixed-dose combinations of LAMAs and LABAs that become available during the study and that are captured in each database will be included.
  Interventions: Drug: Aclidinium bromide/formoterol
- New users of other COPD medication: New users of other COPD medications (tiotropium, other LAMAs, LABA, LABA/ICS, LAMA/LABA), prescribed as recorded in the database.
  Interventions: Drug: Other COPD medication

INTERVENTIONS:
Drug: Aclidinium bromide — Administered as monotherapy, prescribed as recorded in the database.
  Groups: Aclidinium bromide monotherapy
Drug: Aclidinium bromide/formoterol — Administered in combination with formoterol fumarate (concomitant or as a fixed-dose combination), prescribed as recorded in the database.
  Groups: Aclidinium bromide and formoterol
Drug: Other COPD medication — Other COPD medication including:
  tiotropium; other long-acting anticholinergic (LAMAs; lycopyrronium bromide, umeclidinium); LABA (formoterol, salmeterol, indacaterol); LABA/ICS (formoterol/budesonide, formoterol/beclometasone, formoterol/mometasone, formoterol/fluticasone, salmeterol/fluticasone propionate, and vilanterol/fluticasone); LAMA/LABA (approved or under regulatory review or in development; glycopyrrolate/formoterol, glycopyrronium/indacaterol, tiotropium/olodaterol, umeclidinium/vilanterol), prescribed as recorded in the database.
  Groups: New users of other COPD medication

SUMMARY:
DUS1 and DUS2 are descriptive drug utilisation studies in new users of aclidinium bromide in Europe.

The objectives of DUS1 and DUS2 are to describe the characteristics and patterns of use of new users of aclidinium bromide (monotherapy or in combination) and new users of other medications for chronic obstructive pulmonary disease (COPD); to evaluate the potential off-label use of aclidinium bromide; to describe users of aclidinium bromide in subgroups of patients for whom there is missing information in the risk management plan (RMP); and to establish a core cohort of new users of aclidinium bromide for the future evaluation of safety concerns described in the RMP.

The data source for these studies will be the CRPD in the UK, the GePaRD in Germany, and national health databases in Denmark.

DETAILED DESCRIPTION:
DUS1 will be conducted when the target number of new users of aclidinium monotherapy is reached, and DUS2 when the target number of new users of aclidinium fixed-dose combination with formoterol is reached.

As this was a descriptive study no primary or secondary endpoints were specified.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the study will be required to meet the following criteria, as ascertained from each of the automated databases:
* To have at least 1 year of enrolment in the database (DUS1 and DUS2).
* To have not been prescribed aclidinium bromide as monotherapy or with concomitant use of formoterol during the 6 months before the date of first prescription of aclidinium bromide (index date) in DUS1
* To have not been prescribed aclidinium bromide as monotherapy, with concomitant use of formoterol, or as aclidinium/formoterol during the 6 months before the date of first prescription of aclidinium bromide (index date) in DUS2

The same inclusion criteria will be applied for each of the comparator drugs.

Exclusion Criteria:

* No age restrictions or exclusion criteria will be applied. This will allow for the characterisation of all users of aclidinium bromide and comparator drugs irrespective of the indication for which these medications are used. Identification of potential off-label use of aclidinium bromide in the paediatric and adult populations is one of the specific objectives of this DUS.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: New users of aclidinium bromide (on monotherapy or with concomitant use of formoterol) and new users of other COPD medications will be identified and included in the specific exposure cohort of interest.
Sampling Method: Probability Sample
Enrollment: 22155 (Actual)
Dates: Start 2015-07-06 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Baseline age of new users | Baseline (date of first prescription)
Baseline frequency of new users with a diagnosis of COPD including emphysema or chronic bronchitis | Baseline (date of first prescription)
Baseline frequency of new users with severe COPD | Baseline (date of first prescription)
  COPD severity including recent exacerbations
Baseline frequency of new users with a history of cardiovascular disease | Baseline (date of first prescription)
  Baseline history of cardiovascular diseases and baseline cardiovascular risk profile, including diabetes, recent acute myocardial infarction (AMI), unstable angina, arrhythmias, or heart failure
Overall comorbidity index of new users | From date of first prescription up to 1 year of follow-up
Frequency of respiratory medication use by new users | From date of first prescription to 1 year of follow-up
Baseline gender of new users | Baseline (date of first prescription)
Frequency of users of aclidinium bromide with comorbid asthma diagnoses or in the absence of other drugs or diagnoses suggestive of COPD | From date of first prescription up to 1 year of follow-up
Frequency of pregnancies during use of COPD medication | From date of first prescription up to 1 year of follow-up
Frequency of use of aclidinium bromide in the pediatric population | From date of first prescription up to 1 year of follow-up
Frequency of comorbid conditions in the paediatric population | From date of first prescription up to 1 year of follow-up
Baseline frequency of patients with renal or hepatic impairment | Baseline (date of first prescription)
Baseline frequency of patients who have experienced a recent exacerbation | Baseline (date of first prescription
Baseline frequency of patients with thyrotoxicosis or pheochromocytoma | Baseline (date of first prescription)
Frequency of previous smoking in new users | From date of first prescription to 1 year of follow-up
Frequency of current smokers in new users | From date of first prescription to 1 year of follow-up
Frequency of new users with BMI <18.50 kg/m2 (underweight) | From date of first prescription to 1 year of follow-up
Frequency of new users with BMI ranging from 18.50 to 24.99 kg/m2 (normal weight) | From date of first prescription to 1 year of follow-up
Frequency of new users with BMI >25.0 kg/m2 (overweight) | From date of first prescription to 1 year of follow-up
Frequency of new users with BMI ranging between 25.0 and 29.99 kg/m2 (pre-obese) | From date of first prescription to 1 year of follow-up
Frequency of new users with BMI >30 kg/m2 (obese) | From date of first prescription to 1 year of follow-up
Frequency of new users with low socioeconomic status (Townsend multiple deprivation index) | From date of first prescription to 1 year of follow-up
Baseline frequency of patients with benign prostatic hyperplasia | Baseline (date of first prescription)
Baseline frequency of patients with bladder neck obstruction | Baseline (date of first prescription)
Baseline frequency of patients with urinary retention | Baseline (date of first prescription)
Baseline frequency of patients with narrow-angle glaucoma | Baseline (date of first prescription)

SECONDARY OUTCOMES:
Duration of COPD medication use | From date of first prescription up to 1 year of follow-up
  Duration of use will be estimated through the number of consecutive prescriptions, with a maximum interval of 60 days between them, or the days of supply of each prescription, as available in each database.
Average daily dose of COPD medication | From date of first prescription up to 1 year of follow-up
  The daily dose for each treatment will be derived from the recorded dose or from the time between consecutive prescriptions and prescribing information (strength, number of units, and number of boxes) according to the available information in each database.
Adherence to COPD medication within 1 year | From date of first prescription up to 1 year of follow-up
  Consecutive prescriptions are defined as those with a maximum gap of 60 days between the date of prescriptions. Proportion of patients refilling prescriptions within 60 days from the end of the previous prescription.
Frequency of use of concomitant medications | From date of first prescription up to 1 year of follow-up
Frequency of switching between COPD medications | From date of first prescription up to 1 year of follow-up
Total number of prescriptions | From date of first prescription up to 1 year of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Castellsague, MD, MPH, Study Director — RTI Health Solutions; Susana Perez-Gutthann, MD, PhD, Study Director — RTI Health Solutions
Locations (3):
- National Health Database Denmark, Southern Denmark University, Odense, Denmark
- German Pharmacoepidemiological Research Database, Bremen, Germany
- Clinical Practice Research Datalink, London, United Kingdom

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14716&filename=Aclidinium_D6560R00005_(DUS1)_REPORT_SYNOPSIS_20022018.pdf